CLINICAL TRIAL: NCT07357753
Title: Evaluation of the Cancellation of Elective Surgeries on the Day of Operation in Terms of Hospital, Patient, and Cost Outcomes
Brief Title: Evaluation of Same-Day Cancellation of Elective Surgeries
Acronym: DOSCOST
Status: Completed | Type: Observational
Sponsor: Elazıg Fethi Sekin Sehir Hastanesi (Other)
Responsible Party: Principal Investigator, Sevim Şenol Karataş, Principal Investigator, Elazıg Fethi Sekin Sehir Hastanesi
Other Study IDs: FSCH-OR-CANCEL-2025
Record Dates: First submitted 2025-12-18; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Elective Surgery Cancellation; Preoperative Anxiety
Keywords: Elective surgery cancellation; Cancellation reasons; Healthcare costs; Economic impact; Patient anxiety

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cancelled Elective Surgery Cohort: This cohort includes patients whose elective surgical procedures were cancelled on the scheduled day of operation for any reason.

SUMMARY:
This study evaluates elective surgeries that were cancelled on the scheduled day of operation. Same-day surgical cancellations may cause emotional stress for patients, inefficient use of hospital resources, and increased health care costs.

The aim of this observational study is to analyze the reasons for same-day cancellations and to assess their impact on patients, hospital workflow, and costs. Patient anxiety levels after cancellation will be evaluated using standardized questionnaires. The findings of this study may help improve perioperative planning and reduce preventable surgical cancellations.

DETAILED DESCRIPTION:
This prospective observational study was conducted at the operating rooms of Elazığ Fethi Sekin City Hospital. The study included all elective surgical procedures that were cancelled on the scheduled day of operation for any reason after approval by the local ethics committee. Data were collected over a six-month period.

Demographic characteristics of patients, planned surgical procedures, surgical departments, and reasons for cancellation were recorded using patient interviews, medical records, and the hospital information system. Cancellations were categorized as patient-related, hospital-related, or surgery team-related.

The impact of same-day cancellations on hospital resources and costs was evaluated by estimating operating room idle time, personnel costs, unused equipment and medications, bed occupancy, preoperative preparation costs, and additional post-cancellation diagnostic or consultation expenses. Cost calculations were based on official Ministry of Health reimbursement tariffs.

Following cancellation and transfer back to the ward, patients were assessed face to face for anxiety using the State-Trait Anxiety Inventory. The results of this study aim to provide data to improve perioperative planning, optimize hospital resource utilization, and reduce preventable elective surgery cancellations.

This study was registered retrospectively after study completion due to an administrative delay in trial registration.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgical procedures cancelled on the scheduled day of operation for any reason.

Exclusion Criteria:

* Patients who could not be contacted on the day of cancellation.

Patients with insufficient medical or administrative data in their records.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients scheduled for elective surgery whose procedures were cancelled on the scheduled day of operation at Elazığ Fethi Sekin City Hospital
Sampling Method: Non-Probability Sample
Enrollment: 408 (Actual)
Dates: Start 2025-03-25 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-10 (Actual)

PRIMARY OUTCOMES:
Reasons for same-day cancellation of elective surgeries | From the date of scheduled elective surgery to the end of the same calendar day on which the cancellation occurred, assessed retrospectively using hospital medical records and patient interviews over a 12-month study period.
  Categorization of cancellation reasons as patient-related, hospital-related, or surgical team-related based on medical records and patient interviews.
Estimated hospital cost associated with cancelled elective surgeries | Perioperative / Periprocedural
  Total estimated cost including operating room idle time, personnel costs, unused equipment and medications, bed occupancy, preoperative preparation costs, and additional post-cancellation diagnostic or consultation expenses.

SECONDARY OUTCOMES:
State anxiety level after surgical cancellation (STAI-State score) | Within 24 hours after cancellation
  The State Anxiety subscale of the State-Trait Anxiety Inventory (STAI-State) is a validated self-report scale ranging from 20 to 80, with higher scores indicating greater levels of anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Fethi Sekin City Hospital, Elâzığ, Elaziğ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No